CLINICAL TRIAL: NCT00515073
Title: A Phase II Study: Paclitaxel and Pelvic Radiation for Stage I-IIIA Papillary Serous Carcinoma of the Endometrium
Brief Title: Papillary Serous Carcinoma of the Endometrium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID00-418
Record Dates: First submitted 2007-08-09; First posted 2007-08-13 (Estimated); Results first posted 2014-07-03 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-05

CONDITIONS: Endometrial Cancer
Keywords: Endometrial Cancer; Papillary Serous Carcinoma; Pelvic Radiation Therapy; Paclitaxel; Taxol
MeSH Terms: conditions — Endometrial Neoplasms; Cystadenocarcinoma, Serous | interventions — Paclitaxel; Dexamethasone; Cimetidine; Diphenhydramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paclitaxel (Taxol) + Pelvic Radiation (Experimental): Paclitaxel (Taxol) 50 mg/m^2 intravenous (IV) weekly over 1 hour for 5 weeks. Radiation therapy to the pelvis daily for 25 treatments.
  Both radiation therapy and paclitaxel chemotherapy on Day 1 or 2, followed by radiation alone for four days, repeated every week for a total of 5 weeks, giving a total dose of 45 Gy with external beam radiation to pelvis and 5 courses of paclitaxel 50 mg/m^2. Four-six weeks after pelvic radiation completed, 4 additional courses of paclitaxel 135 mg/m^2 alone given every 21 days. Vaginal apex boost given either with last 3 external beam treatments or after external beam radiation completed for additional 3 days. No chemotherapy given with vaginal apex boost.
  Interventions: Drug: Paclitaxel; Radiation: Pelvic Radiation; Drug: Dexamethasone; Drug: Cimetidine; Drug: Diphenhydramine

INTERVENTIONS:
Drug: Paclitaxel — 50 mg/m^2 IV over one hour on Day 1, 8, 15, 22, and 29 during radiation therapy followed by 4 additional courses at 135 mg/m^2 IV over 3 hours every 21 days, 4-6 weeks after pelvic radiation is completed.
  Other Names: Taxol
Radiation: Pelvic Radiation — Radiation therapy to the pelvis daily for 25 treatments. Beginning Day 1 or 2 and given for 5 days for 5 weeks, giving a total dose of 45 Gy with external beam radiation to the pelvis. The vaginal apex boost given either with last 3 external beam treatments or after external beam radiation completed for an additional 3 days depending on patient preference. No chemotherapy given with vaginal apex boost.
Drug: Dexamethasone — 20 mg IV given 30 minutes prior to chemotherapy
Drug: Cimetidine — 300 mg IV given 30 minutes prior to chemotherapy
Drug: Diphenhydramine — 50 mg IV given 30 minutes prior to chemotherapy

SUMMARY:
Primary Objectives:

* To evaluate the results of Paclitaxel and pelvic radiation in pelvic confined papillary serous carcinoma of the endometrium for both local control and overall survival.
* To evaluate the toxicity of Paclitaxel and pelvic radiation.
* To collect and evaluate patients' quality of life/symptom assessment data.

DETAILED DESCRIPTION:
Paclitaxel is designed to block the mechanisms of cell division in cancer cells, which may cause them to die.

If you are found to be eligible to take part in this study, you will begin treatment. You will have radiation treatment to your pelvis (hip area) every day (Monday - Friday) for a total of 25 treatments. Each treatment should take about 20 minutes to complete.

After the radiation treatment, you will receive a type of radiation called a "vaginal cuff boost." The vaginal cuff boost involves a small device being inserted into the vagina to treat the back of the vagina with a high dose of radiation. The applicator is similar to placing a large tampon in the vagina. This internal treatment takes about 30 minutes for each treatment. This is separate from the external radiation treatments that are given.

While you are receiving radiation treatment, and then afterwards, you will also receive chemotherapy with paclitaxel. During the radiation period, you will receive paclitaxel by vein over 1 hour, on Days 1, 8, 15, 22, and 29. Starting 4-6 weeks after radiation treatment is finished, you will receive paclitaxel at a larger dose, given over 3 hours each time, once every 21 days (3 weeks). You will receive up to 4 "cycles" of chemotherapy, each cycle lasting 21 days.

You will be given certain drugs about 30 minutes before your chemotherapy treatments to help control possible side effects, like allergic reactions. These drugs include dexamethasone, diphenhydramine (Benadryl), and cimetidine.

You will have several tests performed throughout the study. Before each cycle of chemotherapy and one month after the last cycle of chemotherapy is given, quality of life and symptom assessment forms will be completed. These questionnaires should only take about 15 minutes to complete.

While you are on chemotherapy treatment, you will have tests performed before each chemotherapy treatment. This will involve blood (about 1 tablespoon) drawn for routine tests, and a review of your symptoms by the study staff.

Once you are off study treatment, you will be asked to return to the clinic for follow-up visits. These visits will occur every 3 months for 1 year, then every 4 months for 2 years, then every 6 months for 2 years, then once a year after that. At these visits, you will have a physical and pelvic exam performed, along with blood (about 1 tablespoon) drawn for routine tests. Chest x-rays will usually be done once a year and any other diagnostic exams will only be done if your doctor thinks they are needed.

This is an investigational study. There are no standard treatments for this type of endometrial cancer, but radiation and chemotherapy are common treatments. This combination of chemotherapy and radiation is considered experimental. Up to 49 patients will take part in this multicenter study. Up to 44 participants will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must undergo surgical staging within 8 weeks of study entry.
2. Patients with mixed histology tumor that include a papillary serous component are eligible.
3. Only patients with non-measurable disease can be entered.
4. Patients may not have had previous chemotherapy or radiation therapy.
5. Patients must have an estimated life expectancy of 12 weeks or greater.
6. Patients must have a Zubrod performance status of less than or equal to 2.
7. Patients must have adequate bone marrow, renal and hepatic function: with white blood count (WBC) greater than or equal to 3000; Absolute neutrophil count (ANC) greater than or equal to 1500; Platelets greater than or equal to 100,000; glutamic-pyruvic transaminase (SGPT) less than or equal to 2 times the upper limit of normal; Total bilirubin less than or equal to 2.5mg/dl.
8. Patients must sign an institutionally approved consent form

Exclusion Criteria:

1. Previously treated papillary serous carcinoma with either chemotherapy or radiation therapy.
2. Newly diagnosed papillary serous carcinoma of the endometrium, Stage IIIB-IV (patients with disease outside the pelvis).
3. Patients who have a history of other malignancy, with the exception of non-melanomatous skin cancer, unless in complete remission and off all therapy for that disease for a minimum of 5 years.
4. Patients with a Zubrod status of 3 or greater.
5. Patients with an active infection.
6. Patients with serious intercurrent medical illness.
7. Patients with a recent (within 6 months) history of congestive heart failure, unstable angina or myocardial infarction.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2001-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anuja Jhingran, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - M. D. Anderson Cancer Center - Orlando, Orlando, Florida
  - UT MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Jhingran A, Ramondetta LM, Bodurka DC, Slomovitz BM, Brown J, Levy LB, Garcia ME, Eifel PJ, Lu KH, Burke TW. A prospective phase II study of chemoradiation followed by adjuvant chemotherapy for FIGO stage I-IIIA (1988) uterine papillary serous carcinoma of the endometrium. Gynecol Oncol. 2013 May;129(2):304-9. doi: 10.1016/j.ygyno.2013.01.025. Epub 2013 Feb 4. PMID 23385150
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: April 30, 2001 to November 18, 2009 with actual enrollment occuring October 2001 through July 2009 at University of Texas (UT) MD Anderson Cancer Center and MD Anderson Cancer Center Orlando.
Pre-assignment Details: Two participants of 32 were enrolled but not included in group assignment due to ineligibility.
Groups:
- Paclitaxel (Taxol) + Pelvic Radiation: Paclitaxel (Taxol) 50 mg/m^2 intravenous (IV) weekly over 1 hour for 5 weeks. Radiation therapy to the pelvis daily for 25 treatments.
  Both radiation therapy and paclitaxel chemotherapy on Day 1 or 2, followed by radiation alone for four days, repeated every week for a total of 5 weeks, giving a total dose of 45 Gy with external beam radiation to pelvis and 5 courses of paclitaxel 50 mg/m^2. Four-six weeks after pelvic radiation completed, 4 additional courses of paclitaxel 135 mg/m^2 alone given every 21 days. Vaginal apex boost given either with last 3 external beam treatments or after external beam radiation completed for additional 3 days. No chemotherapy given with vaginal apex boost.
  Dexamethasone 20 mg, Diphenhydramine 50 mg and Cimetidine 300 mg IV 30 minutes prior to chemotherapy.
Period: Overall Study
Arm/Group | Paclitaxel (Taxol) + Pelvic Radiation
Started | 30
Completed | 28
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Paclitaxel (Taxol) + Pelvic Radiation
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 63 [36 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival at 2 Years and 5 Years
Description: The percentage of participants who are still alive for A designated period of time (2 years and 5 years) after starting treatment. Continual Assessments every 3 months for 1 year, then every 4 months for 2 years, then every 6 months for 2 years, then once a year.
Time Frame: Assessment at 2 years and 5 years
Population: Two participants were inevaluable.
Measure: Number; unit: percentage of participants
Arm/Group | Paclitaxel (Taxol) + Pelvic Radiation
Number analyzed (Participants) | 28
percentage of participants
  2 Years | 93
  5 Years | 85

ADVERSE EVENTS:
Time Frame: Adverse events elicited at each clinic visit during participation in the study, approximately 15 weeks of treatment with 2 year follow up. Overall study period from November 2001 to December 2009.
Arm/Group | Paclitaxel (Taxol) + Pelvic Radiation
Serious Adverse Events (participants affected / at risk) | 15/30
Other Adverse Events (participants affected / at risk) | 19/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel (Taxol) + Pelvic Radiation (N=30)
GRANULOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1)
FATIGUE (General disorders) | 10 (10)
NAUSEA (Gastrointestinal disorders) | 5 (5)
VOMITING (Gastrointestinal disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 13 (13)
PAIN, ABDOMEN (General disorders) | 2 (2)
HEADACHE (Nervous system disorders) | 2 (2)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 6 (7)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (2)
ANXIETY (Psychiatric disorders) | 1 (1)
PAIN, CHEST (General disorders) | 1 (1)
PAIN, BONE (Musculoskeletal and connective tissue disorders) | 3 (3)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1)
INFECTION (Infections and infestations) | 2 (2)
ANOREXA (Metabolism and nutrition disorders) | 5 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel (Taxol) + Pelvic Radiation (N=30)
CONSTIPATION (Gastrointestinal disorders) | 2 (3)
DIAPHORESIS (Skin and subcutaneous tissue disorders) | 3 (3) — Sweating
DIARRHEA (Gastrointestinal disorders) | 8 (12)
FATIGUE (General disorders) | 7 (9)
FEVER WITHOUT NEUTROPENIA (Investigations) | 2 (2)
GLUCOSE, SERUM-HIGH (Metabolism and nutrition disorders) | 2 (2)
GRANULOCYTOPENIA (Blood and lymphatic system disorders) | 3 (3)
HEADACHE (Nervous system disorders) | 4 (4)
HYPOKALEMIA (Metabolism and nutrition disorders) | 4 (4)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 2 (2)
LEUKOPENIA (Blood and lymphatic system disorders) | 9 (9)
MOTOR SKILL (Musculoskeletal and connective tissue disorders) | 4 (4)
MUCOSITIS (CLINICAL EXAM) ORAL CAVITY (Gastrointestinal disorders) | 2 (2)
MYALGIA (General disorders) | 5 (11)
NAUSEA (Gastrointestinal disorders) | 3 (7)
PAIN (ABDOMEN NOS) (General disorders) | 2 (6)
PAIN (General disorders) | 2 (2) — Bone, Extremity-Limb
RIGORS, CHILLS (General disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (5)
NEUROPATHY (Nervous system disorders) | 16 (16)
ANOREXIA (Gastrointestinal disorders) | 4 (4)
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 (2)
ANEMIA (Blood and lymphatic system disorders) | 9 (9)
RECTAL BLEEDING (Gastrointestinal disorders) | 2 (2)
INFECTION (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No